CLINICAL TRIAL: NCT04001309
Title: A Randomized Antimicrobial Stewardship Trial in a Hospital Setting
Brief Title: Antimicrobial Stewardship Interventions in a Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Thomas Tängdén, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2018-423
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Infectious Disease
Keywords: antimicrobial stewardship; prospective audit and feedback; infectious diseases; randomized trial
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Masking for care providers and investigators is not feasible. Outcomes assessors will be blinded to study period and intervention arms when evaluating appropriateness of prescribing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infectious diseases physician led (Experimental): Prospective audit and feedback of antimicrobial therapy by infectious disease physicians twice weekly
  Also including standard of care
  * infectious disease consultant on demand
  * hospital antimicrobial stewardship program as usual (education, general information, feedback on prescribing)
  Interventions: Other: Implementation of prospective audit and feedback stewardship interventions to reduce unnecessary use of antimicrobials and improve quality of prescriptions
- Multiprofessional team (Experimental): Prospective audit and feedback of antimicrobial therapy by infectious disease physicians once weekly, ward clinical pharmacists thrice weekly and engagement of ward nurses in the stewardship intervention
  Also including standard of care
  * infectious disease consultant on demand
  * hospital antimicrobial stewardship program as usual (education, general information, feedback on prescribing)
  Interventions: Other: Implementation of prospective audit and feedback stewardship interventions to reduce unnecessary use of antimicrobials and improve quality of prescriptions

INTERVENTIONS:
Other: Implementation of prospective audit and feedback stewardship interventions to reduce unnecessary use of antimicrobials and improve quality of prescriptions — Prospective audit and feedback of antimicrobial therapy at hospital wards, by interventions performed by infectious diseases specialists alone or using a team-based approach.

SUMMARY:
The emerging crisis of multidrug-resistant bacteria is accelerated by a massive overuse and misuse of antibiotics. It has been estimated that 50% of antibiotic prescriptions are inappropriate. Antibiotic interventions to improve prescribing patterns have been successfully implemented in primary care in Sweden and other countries. However, much of the last-resort antibiotics are used in hospitals in which decisions on therapy for bacterial infections are more complex. In this project we will explore the appropriateness of antibiotic prescribing in a hospital setting and measures to improve the quality of antimicrobial therapy. Antimicrobial stewardship interventions will be conducted at selected hospital departments using prospective audit and feedback in a multifaceted and cross-disciplinary approach. The intervention effects on antibiotic consumption, appropriateness of prescriptions, patient outcome and emergence of resistance will be evaluated, and a financial cost-effectiveness analysis will be performed.

DETAILED DESCRIPTION:
Background: In this project we will address the issue of inappropriate antibiotic prescribing in a hospital setting using a systematic and cross-disciplinary approach. We believe that a substantial reduction in antibiotic use and a significant improvement in prescribing patterns can be achieved, which will benefit the patients by reducing the risks of side effects such as antibiotic-induced Clostridium difficile enteritis.

Aim: The aim of this study is to implement and evaluate antibiotic interventions at targeted hospital wards.

Method: Hospital wards will be randomised to one of two antimicrobial stewardship intervention arms stratified by specialty (medicine or surgery). Prospective audit and feedback is a core intervention strategy in both arms.

Statistics: Interrupted time-series analysis (ITS) will be used for the primary endpoint; volume of antimicrobial prescribing. Monthly baseline data at least five years prior to start of the intervention and a during a follow-up period of at least 12 months after end of the intervention period will be used to assess immediate and sustained effects.

Endpoints and outcomes:

* Primary endpoint is reduction in antibiotic use, days of antibiotic therapy (DOTs)/100 patient days
* Secondary endpoints include outcome measures for quantity of antibiotic use, appropriateness of prescriptions, clinical and microbiological outcome and cost-effectiveness.

Data on antibiotic use and trends in prescriptions of key antibiotics will be obtained from hospital pharmacies. Data on duration of hospitalization, patient mortality, re-admissions and side effects including antibiotic-associated Clostridium difficile enteritis will be extracted from the medical records to assess potential impact on patient outcome caused by the intervention. Data on emergence of resistance during therapy and general trends in resistance epidemiology will be recorded. The outcome assessment will include a survey to participating physicians on the value different aspects of the stewardship intervention in their daily care of patients with infections. A cost-effectiveness analysis of the intervention will be performed.

ELIGIBILITY:
Randomization to intervention arms is performed on ward level.

Eligibility criteria:

- Surgical or medical wards

Patient level (too be included in the outcome analyses)

Inclusion Criteria:

* At least 18 years of age
* Ongoing antimicrobial therapy on a study ward
* Signed informed consent

Exclusion Criteria:

* Patients in palliative care with very short life expectancy
* Patients from another county than study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change and trends in days of antibiotic therapy (DOT)/100 patient days | 7 years
  Monthly DOT of antibiotics per 100 patient days on ward level assessed 5 y pre-intervention and 1 y post-intervention. Data will be analysed using interrupted time series analysis to assess immediate changes following implementation and comparison of trends before and after the intervention.

SECONDARY OUTCOMES:
Days of defined daily doses (DDDs)/100 patient days | 12 months
  Overall days of therapy per 100 patient days (PD) on the ward level
Treatment duration (Days per treatment period overall) | 12 months
  Overall days per treatment episode. A treatment episode is defined as antimicrobial treatment not interrupted by more than one calendar day.
30-d mortality | 12 months
  All cause 30-d mortality
In-hospital mortality | 12 months
  All-cause in-hospital mortality
Hospital readmission within 30 d after discharge | 12 months
  Unplanned hospital readmission within 30 d after discharge
Hospital readmission due to relapse of infection within 30 d after discharge | 12 months
  Unplanned hospital readmission due to relapse of infection within 30 d after discharge
Hospital length of stay (LOS) | 12 months
  Hospital length of stay per admission
Intensive Care Unit (ICU) transfer | 12 months
  Proportion of admissions transferred to ICU after initial non-ICU admission
Guideline compliance | 12 months
  Proportion of patients treated where antimicrobial therapy was in compliance with local guideline, or in absence of local guideline national guideline
De-escalation or shift to targeted therapy | 12 months
  Proportion of patients where de-escalation or shift to targeted antibiotic therapy occurred within 72 hours after initiation of treatment
Intravenous to oral switch | 12 months
  Proportion of patients where intravenous antibiotics was shifted to oral therapy within 5 days (if appropriate)
Appropriate diagnostic examinations | 12 months
  Proportion of patients with appropriate diagnostic examinations performed, according to local guidelines, or in the absence of local guidelines national guidelines
Dose adjustment for renal function within 48 h after initiation of antimicrobial therapy at admission | 12 months
  Dose adjustment of antimicrobial after the most critical phase of the infection
Dose adjustment for renal function when initiating antimicrobial therapy in a non-acute situation | 12 months
  Proportion of antimicrobial prescription in non-acute situations where dosing was according to renal function
Therapeutic drug monitoring (TDM) | 12 months
  Proportion of patients where TDM was used, when applicable according to local guideline
Drug-drug interactions (DDI) | 12 months
  Important DDI taken into account when prescribing antimicrobial therapy
Incidence of Clostridium difficile infections (CDI) | 12 months
  Incidence of healthcare-facility onset CDI denominated by 10 000 PD and admission
Incidence of multidrug-resistant organisms (MDRO) | 12 months
  Incidence of clinical cultures with multidrug resistant organisms (methicillin-resistant Staphylococcus aureus (MRSA), Extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E), carbapenemase-producing Enterobacteriaceae (CPE), vancomycin-resistant enterococci (VRE), multidrug resistant P. aeruginosa) denominated per 1000 PD and admissions
Costs of administered antimicrobials | 12 months
  Costs of administered antimicrobials (overall and by class) per admission and per patient receiving antibiotics
Costs of the intervention | 12 months
  Total costs of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tängdén, MD, Phd, Principal Investigator — Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Uppsala University Hospital, Uppsala
  - Ystads lasarett, Ystad